CLINICAL TRIAL: NCT01615354
Title: Single-Center, Randomized, Double-Blind, Placebo Controlled, Crossover Study to Assess the Effect of Aleglitazar on the Pharmacokinetics and Pharmacodynamics of Ethinyl Estradiol and Levonorgestrel as Components of the Oral Contraceptive Microgynon®
Brief Title: A Study of Aleglitazar in Combination With Oral Contraceptive Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: BP25559
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — aleglitazar; ethinyl estradiol, levonorgestrel drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Microgynon®; Drug: Placebo
- Treatment (Experimental)
  Interventions: Drug: Aleglitazar; Drug: Microgynon®

INTERVENTIONS:
Drug: Aleglitazar — Multiple oral doses
  Arms: Treatment
Drug: Microgynon® — Multiple oral doses
Drug: Placebo — Multiple oral doses
  Arms: Placebo

SUMMARY:
This randomized, double-blind, placebo-controlled, cross-over study will assess the effect of aleglitazar on the pharmacokinetics and pharmacodynamics on Microgynon® in healthy volunteers. Volunteers will receive multiple oral doses of aleglitazar in one period; in the other period volunteers will receive placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteer, 18 to 45 years of age
* Body mass index (BMI) between 18.0 and 29.9 kg/m2
* Body weight at least 55.0 kg
* Non-pregnant, not lactating and not planning pregnancy from screening to 3 months after the last dose of study treatment
* Non-smoker for at least 3 months

Exclusion Criteria:

* Currently active gynecological disorder
* History of amenorrhea within the previous 3 years
* Known or suspected history of estrogen-dependent neoplasia or sex hormone-dependent malignant tumors
* Use of steroid hormone-containing intrauterine device (IUD) or progesterone-release IUD contraceptive within 3 months to screening.
* History of clinically significant disease that could jeopardize the volunteer safety in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of Levonorgestrel: area under the concentration time curve | pre-dose and up to 24 hours post-dose
Pharmacokinetics of ethinyl estradiol: area under the concentration time curve | pre-dose and up to 24 hours post-dose

SECONDARY OUTCOMES:
Pharmacodynamics: luteinizing/follicular stimulation hormone concentration | Days 1, 7, 13, 14, 15, 21
Safety: incidence of adverse events | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Manchester, United Kingdom